CLINICAL TRIAL: NCT01885013
Title: Phase II Comparative Study of Myocet Plus Cyclophosphamide in First Line Treatment of HER2 Negative Metastatic Breast Patients
Brief Title: Myocet + Cyclophosphamide + Metformin Vs Myocet + Cyclophosphamide in 1st Line Treatment of HER2 Neg. Metastatic Breast Cancer Patients
Acronym: MYME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRST174.04; 2009-014662-26 (EudraCT Number)
Record Dates: First submitted 2013-06-19; First posted 2013-06-24 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Human Epidermal Growth Factor 2 Negative Carcinoma of Breast
Keywords: HER2 negative; metastatic breast cancer; non endocrine responsive disease
MeSH Terms: conditions — Breast Neoplasms | interventions — Metformin; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin + Myocet + Cyclophosphamide (Experimental): arm A : Metformin 1000 mg, 2 times daily per os*. Myocet 60 mg/m2, intravenous infusion, on day 1, every 21 days Cyclophosphamide 600 mg/m2, intravenous infusion, at day 1 every 21 days.
  * During cycle 1, patients will assume only metformin from day 1 to day 13 and will begin chemotherapy from day 14. From day 1 to day 3, patients will assume Metformin 1000 mg once a day. Starting from day 4 patients will assume Metformin 1000 mg 2 times a day.
  Interventions: Drug: Metformin + Myocet + Cyclophosphamide
- Myocet + Cyclophosphamide (Active Comparator): arm B : Myocet 60 mg/m2, intravenous infusion, on day 1, every 21 days Cyclophosphamide 600 mg/m2, intravenous infusion, on day 1, every 21 days
  Interventions: Drug: Myocet + Cyclophosphamide

INTERVENTIONS:
Drug: Metformin + Myocet + Cyclophosphamide — Metformin + Myocet + Cyclophosphamide:
  Metformin 1000 mg, 2 times daily per os*. Myocet 60 mg/m2, intravenous infusion, on day 1, every 21 days Chemotherapy will be performed for 8 cycles Cyclophosphamide 600 mg/m2, intravenous infusion, at day 1 every 21 days.
  * During cycle 1, patients will assume only metformin from day 1 to day 13 and will begin chemotherapy from day 14. From day 1 to day 3, patients will assume Metformin 1000 mg once a day. Starting from day 4 patients will assume Metformin 1000 mg 2 times a day.
  Other Names: metformin; myocet; cyclofosfamide
  Arms: Metformin + Myocet + Cyclophosphamide
Drug: Myocet + Cyclophosphamide — Myocet + Cyclophosphamide:
  Myocet 60 mg/m2, intravenous infusion, on day 1, every 21 days Cyclophosphamide 600 mg/m2, intravenous infusion, on day 1, every 21 days Chemotherapy will be performed for 8 cycles
  Other Names: myocet; cyclofosfamide
  Arms: Myocet + Cyclophosphamide

SUMMARY:
This is a phase II comparative randomized clinical trial.

Eligible patients will be randomized (1:1) to:

Arm A: Myocet plus Cyclofosfamide plus Metformin Arm B: Myocet plus Cyclofosfamide

Statistical Considerations:

In this randomized phase II study, the sample size was calculated basing on the primary end-point (PFS) and assuming an error α = 10% (2-tailed) with a power of 80%.

To find an advantage of 4 months of median time to progression (6 months in the control arm B and 10 months in the experimental arm A) will be recruited 112 patients (98 events) for a period of 24 months and will be considered further 12-month of follow-up. The primary analysis of the study will be conducted in accordance with the "intention to treat" principle, the secondary analysis will be conducted in the "per protocol" population.

DETAILED DESCRIPTION:
MULTICENTER, RANDOMIZED, COMPARATIVE STUDY OF MYOCET PLUS CYCLOPHOSPHAMIDE PLUS METFORMIN VERSUS MYOCET PLUS CYCLOPHOSPHAMIDE IN FIRST LINE TREATMENT OF HER2 NEGATIVE METASTATIC BREAST CANCER PATIENTS.

The aim of this study is to determine if the addition of metformin to the regime Myocet / Cyclophosphamide improves disease-free survival in patients with HER2-negative metastatic breast cancer.

The primary objective is the evaluation of the clinical efficacy of the combination of Myocet / Cyclophosphamide plus Metformin compared to treatment with only Myocet / Cyclophosphamide, in terms of progression-free survival (PFS).

Clinical secondary objectives are:

* Objective response rate
* Overall survival
* Tolerability
* Progression-free survival, objective response rate and overall survival according to Homa Index levels.

Secondary biological endpoint is the characterization of the metabolic profile of patients (sensitivity in insulin levels).

Treatment Arm A (experimental treatment):

Metformin 1000 mg, 2 times daily per os*. Myocet 60 mg/m2, intravenous infusion, on day 1, every 21 days Cyclophosphamide 600 mg/m2, intravenous infusion, at day 1 every 21 days.

* During cycle 1, patients will assume only metformin from day 1 to day 13 and will begin chemotherapy from day 14. From day 1 to day 3, patients will assume Metformin 1000 mg once a day. Starting from day 4 patients will assume Metformin 1000 mg 2 times a day.

Arm B (standard treatment):

Myocet 60 mg/m2, intravenous infusion, on day 1, every 21 days Cyclophosphamide 600 mg/m2, intravenous infusion, on day 1, every 21 days

Chemotherapy will be performed for 8 cycles.

The treatment will be continued until progression of disease.

Statistical Considerations:

In this randomized phase II study, the sample size was calculated basing on the primary end-point (PFS) and assuming an error α = 10% (2-tailed) with a power of 80%.

To find an advantage of 4 months of median time to progression (6 months in the control arm B and 10 months in the experimental arm A) will be recruited 112 patients (98 events) for a period of 24 months and will be considered further 12-month of follow-up. The primary analysis of the study will be conducted in accordance with the "intention to treat" principle, the secondary analysis will be conducted in the "per protocol" population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed breast cancer
2. Metastatic disease
3. HER2 negative disease, as measured by IHC or FISH
4. Non endocrine responsive disease (negative hormonal status or failure of endocrine therapy for MBC)
5. Patients with measurable and/or non-measurable disease according to RECIST Criteria (Version 1.1)
6. Homa Index calculated according to Matthews' formula
7. Prior endocrine therapy is allowed, in the adjuvant and/or metastatic setting
8. Prior chemotherapy is allowed, only in adjuvant setting, provided it is terminated at least 12 months before study entry. Adjuvant anthracyclines are allowed if prior cumulative dose does not exceed 360 mg/m2 in case of epirubicin and 280 mg/m2 in case of doxorubicin. Adjuvant taxanes are allowed.
9. Age 18-75 years
10. Life expectancy of greater than 3 months
11. ECOG performance status <2
12. Patients must have normal organ and marrow function:

    * leukocytes >=3,000/μL
    * absolute neutrophil count >=1,500/μL
    * platelets >=100,000/μL
    * total bilirubin within normal institutional limits
    * AST(SGOT)/ALT(SGPT) <=1.5 X institutional upper limit of normal
    * creatinine within normal institutional limits
13. Adequate cardiac function, i.e. left ventricular ejection fraction (LVEF)>= 50%
14. The effects of liposomal doxorubicin on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because anthracyclines as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. All women of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to the start of study medication. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
15. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Known diabetes (type 1 or 2)
2. Currently on metformin, sulfonylureas, thiazolidenediones or insulin for any reason (these drugs alter insulin levels)
3. Current or previous congestive heart failure, renal failure or liver failure; history of acidosis of any type; habitual intake of 3 or more alcoholic beverages per day
4. Creatinine above upper limit of normal for institution, AST above 1.5 times upper limit or normal for institution (to reduce risk of lactic acidosis)
5. Hypersensitivity or allergy to metformin
6. Participation in another clinical trial with any investigational agents within 30 days prior to study screening
7. Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
8. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Myocet or other agents used in the study
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2010-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 42 months
  Clinical efficacy of the combination of Myocet / Cyclophosphamide plus Metformin compared to treatment with only Myocet / Cyclophosphamide, in terms of progression-free survival (PFS)

SECONDARY OUTCOMES:
Objective response rate | 42 months
  Objective Response Rate after treatment with Myocet/Cyclophosphamide/Metformin compared with after therapy with Myocet/Cyclophosphamide
Overall survival | 42 months
  Overall survival after treatment with Myocet/Cyclophosphamide/Metformin compared with after therapy with Myocet/Cyclophosphamide
Progression free survival as function of Homa Index levels | 42 months
  Clinical efficacy of the combination of Myocet / Cyclophosphamide plus Metformin compared to treatment with only Myocet / Cyclophosphamide, in terms of progression-free survival (PFS) as function of Homa Index levels
objective response rate as function of Homa Index levels | 42 months
  Objective Response Rate after treatment with Myocet/Cyclophosphamide/Metformin compared with after therapy with Myocet/Cyclophosphamide, as function of Homa Index levels
overall survival as function of Homa Index levels | 42 months
  Overall survival after treatment with Myocet/Cyclophosphamide/Metformin compared with after therapy with Myocet/Cyclophosphamide, as function of Homa Index levels
patient metabolic profile (metabolic syndrome) | 42 months
  Characterization of the metabolic profile of patients: sensitivity in insulin levels

CONTACTS AND LOCATIONS:
Overall Officials: Dino Amadori, MD, Principal Investigator — IRST IRCCS, Meldola
Locations (25):
- Italy (25):
  - P.O. M. Bufalini, Cesena, FC
  - UO Oncologia Medica IRCCS IRST, Meldola (FC), FC
  - Ospedale Civile degli Infermi, Faenza, RA
  - Ospedale Umberto I, Lugo, RA
  - Ospedale Civile Santa Maria delle Croci, Ravenna, RA
  - ULSS n.8 Asolo Ospedale di Castelfranco, Asolo
  - Centro di Riferimento Oncologico CRO, Aviano
  - Ospedale S.Martino, Belluno
  - Azienda Ospedaliera "Antonio Cardarelli", Campobasso
  - P.O. "SS. Annunziata", Chieti
  - Presidio Ospedaliero E. Profili, Fabriano
  - E.O. Galliera, Genova
  - Ospedale di Guastalla, Guastalla
  - Azienda per i Servizi Sanitari n.5 "Bassa Friulana", Latisana
  - Presidio Ospedaliero "Vito Fazzi", Lecce
  - ULSS n.13 di Mirano, Mirano
  - Arcispedale S. Maria Nuova, Modena
  - Azienda Ospedaliera S. Salvatore di Pesaro, Pesaro
  - Ospedale S. Spirito, Pescara
  - Ospedale Civile di Piacenza, Piacenza
  - Azienda Ospedaliera Santa Maria degli Angeli, Pordenone
  - Arcispedale S. Maria Nuova, Reggio Emilia
  - Ospedale Civile degli Infermi, Rimini
  - IRCCS Centro di riferimento Oncologico di Basilicata di Rionero in Vulture, Rionero in Vulture
  - Ospedale Nuovo Regina Margherita, Roma

REFERENCES:
- [Derived] Gennari A, Foca F, Zamarchi R, Rocca A, Amadori D, De Censi A, Bologna A, Cavanna L, Gianni L, Scaltriti L, Rossi E, Facchinetti A, Martini V, Bruzzi P, Nanni O. Insulin-like growth factor-1 receptor (IGF-1R) expression on circulating tumor cells (CTCs) and metastatic breast cancer outcome: results from the TransMYME trial. Breast Cancer Res Treat. 2020 May;181(1):61-68. doi: 10.1007/s10549-020-05596-4. Epub 2020 Mar 21. PMID 32200486